CLINICAL TRIAL: NCT03940755
Title: Long-term Outcomes of Critical Illness Survivors：a Prospective Cohort Study
Brief Title: Long-term Outcomes of Critical Illness Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jian-jun Yang (Other)
Responsible Party: Sponsor-Investigator, Jian-jun Yang, Director,Department of Anesthesiology, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Other Study IDs: 20190501
Record Dates: First submitted 2019-05-01; First posted 2019-05-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Intensive Care Units

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critical Illness Survivors: Those intensive care unit(ICU) patients who survive from critical illness.

SUMMARY:
The goal of this study is to assess the Long-term Outcomes of Critical Illness Survivors,including physical, psychological, and cognitive sequelae.

DETAILED DESCRIPTION:
An increasing number of patients survive critical illness; however, the evidence reveals that over the same period the number of patients being sent to rehabilitation settings have tripled . For those who do survive, the latest data indicate that 50-70% of ICU "survivors" will suffer cognitive impairment and 60-80% of "survivors" will suffer functional impairment or ICU-acquired weakness (ICU-AW).Still,there is a lack valid data on the long-term impact on morbidity from prospective observational studies. Therefore, the investigators designed an observational cohort which cover a broader range of outcomes to quantify long-term physical, psychological, and cognitive impairment after intensive care unit (ICU).Intensive Care Unit patients survive from critical illness will be approached for study recruitment and participation.Survival rate,Quality of life,Cognitive impairments,Depression and anxiety,PTSD,Physical activity,Neuromuscular impairment will be assessed 3 or 6 months after ICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >17 years
* Patients in intensive care unit(ICU) with at least one organ or system dysfunction,such as respiratory failure, cardiogenic shock,or septic shock.

Exclusion Criteria:

* Refuse to participate
* Death before ICU discharge
* pre-existing cognitive impairment, malignant tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients of Jiangyin people's hospital
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Survival rate of ICU survivors | 3 or 6 months after ICU discharge
  Critically ill patients discharged from ICU are defined as survivors

SECONDARY OUTCOMES:
Assessment of life quality | 3 or 6 months after ICU discharge
  Quality of Life assessed with help of The 36-item short from health survey(SF-36)questionnaire.The SF-36 has 8 scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0-100. Lower scores = more disability, higher scores = less disability.The 8 sections are listed below:PF：Physical Functioning,RP：Role-Physical,BP：Bodily Pain,GH:General Health,VT：Vitality,SF：Social Functioning,RE：Role-Emotional,MH：Mental Health.
Assessment in Physical dysfunction | 3 or 6 months after ICU discharge
  Functional disabilities assessed with help of Barthel index of ADL(activities of daily living).10 variables are addressed. Range of summed total score: 0-100. higher values represent better outcome.
Assessment in depression and anxiety | 3 or 6 months after ICU discharge
  Depression and anxiety assessed with help of The Hospital Anxiety and Depression Scale(HADS).For Depression(D), 7 questions in total. Range of score for each question: 0-3. Total score summed: 0-21 ;For Anxiety(A): 7 questions in total. Range of score for each question: 0-3. Total score summed: 0-21 .For both D and A scales, higher scores represent worse outcome.
Assessment in PTSD | 3 or 6 months after ICU discharge
  Post-traumatic stress syndrome assessed with help of trauma screening questionnaire(TSQ).There are 10 questions in the TSQ. For each question, the answer is either YES or NO. More YES = worse outcome. At least 6 YES represents PTSD diagnosis.
Assessment in Cognitive impairments | 3 or 6 months after ICU discharge
  Cognitive impairments assessed with help of mini-mental state examination(MMSE).The MMSE has 5 scaled scores; the scores are weighted sums of the questions in each section. The 5 sections and their range of score are listed below:Orientation 0-10;Registration 0-3;Attention and calculation 0-5;Recall 0-3;Language 0-9.Total score range from 0-30. Lower scores = more disability, higher scores = less disability.
Patients' care and support needs;social and economical consequences | 3 or 6 months after ICU discharge
  Patients' information of specific needs and supports and social or economical impact post ICU.
Neuromuscular impairment | 3 or 6 months after ICU discharge
  Neuromuscular impairment will be assessed by electromyography/nerve conduction study

CONTACTS AND LOCATIONS:
Overall Officials: Jian-jun Yang, PhD, Principal Investigator — Zhongda Hospital
Locations (2):
- China (2):
  - Jiangyin People's Hospital, Jiangyin, Jiangsu
  - Zhongda Hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] Wischmeyer PE, San-Millan I. Winning the war against ICU-acquired weakness: new innovations in nutrition and exercise physiology. Crit Care. 2015;19 Suppl 3(Suppl 3):S6. doi: 10.1186/cc14724. Epub 2015 Dec 18. PMID 26728966
- [Background] McNelly AS, Rawal J, Shrikrishna D, Hopkinson NS, Moxham J, Harridge SD, Hart N, Montgomery HE, Puthucheary ZA. An Exploratory Study of Long-Term Outcome Measures in Critical Illness Survivors: Construct Validity of Physical Activity, Frailty, and Health-Related Quality of Life Measures. Crit Care Med. 2016 Jun;44(6):e362-9. doi: 10.1097/CCM.0000000000001645. PMID 26974547